CLINICAL TRIAL: NCT00333658
Title: A Behavioral Intervention to Improve Outcomes in VA Work Programs
Brief Title: A Behavioral Intervention to Improve Work Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Bell, Morris - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3108R; MDB0007
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Mental Disorders
Keywords: psychotherapy, group; rehabilitation, vocational; treatment outcome
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intervention
  Interventions: Behavioral: Goal setting and work feedback group
- 2 (No Intervention): Work Services

INTERVENTIONS:
Behavioral: Goal setting and work feedback group — Goal setting and feedback using WBI
  Arms: 1

SUMMARY:
This research has been designed to learn whether getting regular and specific feedback about work performance with small rewards for meeting goals helps people to improve their job performance and leads to better work outcomes, improved mental functioning, and better quality of life

DETAILED DESCRIPTION:
This study is designed to test whether systematic work performance feedback with weekly goal setting, combined with small rewards given for goal achievement, leads to improved vocational, health, and quality of life outcomes for veterans enrolled in the various work service programs at this medical center. The long-term goal of this project is to determine the effectiveness of these interventions at this medical center and to use this experience for a multi-site cooperative study proposal.

Research Design and Methods: One hundred and fifty subjects accepted into work services at this medical center will be randomly assigned to one of two conditions: Work Feedback with Small Rewards, or Usual Services. In the Work Feedback with Small Rewards condition, participants attend a weekly workers meeting where they receive specific feedback based upon the Work Behavior Inventory and set weekly goals. They also receive small rewards for goal achievement that equal $10 per month. Participants in the Usual Services condition do not get specific work feedback but receive all the usual work services normally provided. They also receive $10 per month for active participation. Assessments include baseline evaluations of mental and physical health, social function, cognitive function, and quality of life. Evaluations of mental health, quality of life, and job satisfaction will occur at two months and four months. Six-month and twelve month evaluations will repeat the baseline assessment. Outcome measures will include biweekly work performance assessments, vocational outcomes, mental and physical health status, social and cognitive function, and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Veterans participating in a work program at the VA Connecticut Healthcare System; English-speaking

Exclusion Criteria:

* No exclusion criteria based upon diagnosis, although VA work programs have pre-existing requirements such as a demonstrated need for services, a referral from a clinician, and an interest in work rehabilitation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2003-12; Primary Completion 2007-10 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Competitive employment- | 6 month and 12 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Morris D Bell, PhD, Principal Investigator — VA Connecticut Health Care System (West Haven)
Locations (1):
- VA Connecticut Health Care System (West Haven), West Haven, Connecticut, United States

REFERENCES:
- [Result] Bell MD, Bryson G. Work rehabilitation in schizophrenia: does cognitive impairment limit improvement? Schizophr Bull. 2001;27(2):269-79. doi: 10.1093/oxfordjournals.schbul.a006873. PMID 11354594
- [Result] Bryson G, Bell MD. Initial and final work performance in schizophrenia: cognitive and symptom predictors. J Nerv Ment Dis. 2003 Feb;191(2):87-92. doi: 10.1097/01.NMD.0000050937.06332.3C. PMID 12586961
- [Result] Bell MD, Fiszdon JM, Greig TC, Bryson GJ. Can older people with schizophrenia benefit from work rehabilitation? J Nerv Ment Dis. 2005 May;193(5):293-301. doi: 10.1097/01.nmd.0000161688.47164.71. PMID 15870612